CLINICAL TRIAL: NCT01940393
Title: Evaluation of the Inhibitory Effect of 5 Anti-Histamines in Urticaria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Grupo de Alergología Clínica y Experimental (Other)
Responsible Party: Principal Investigator, Jorge Sanchez, M.D, M.Sc, Allergist, Grupo de Alergología Clínica y Experimental
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GACE-01
Record Dates: First submitted 2013-08-26; First posted 2013-09-12 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Urticaria
Keywords: urticaria; bilastine; fexofenadine; cetirizine; ebastine; desloratadine
MeSH Terms: conditions — Urticaria | interventions — Cetirizine; desloratadine; fexofenadine; ebastine; bilastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cetirizine (Active Comparator): Cetirizine
  Interventions: Drug: Cetirizine
- Desloratadine (Active Comparator): desloratadine
  Interventions: Drug: Desloratadine
- Fexofenadine (Active Comparator): Fexofenadine
  Interventions: Drug: Fexofenadine
- Ebastine (Active Comparator): ebastine
  Interventions: Drug: Ebastine
- Bilastine (Active Comparator): bilastine
  Interventions: Drug: Bilastine

INTERVENTIONS:
Drug: Cetirizine — Drug administration
  Other Names: Alercet
  Arms: Cetirizine
Drug: Desloratadine — Drug Administration
  Other Names: Aerius
  Arms: Desloratadine
Drug: Fexofenadine — Drug administration
  Other Names: Allegra
  Arms: Fexofenadine
Drug: Ebastine — Drug administration
  Other Names: Pinaval
  Arms: Ebastine
Drug: Bilastine — Drug administration
  Other Names: Bilaxten
  Arms: Bilastine

SUMMARY:
The antihistamines with inhaled steroids are the cornerstone on the symptomatic therapy in the management of patients with rhinitis and the first line of treatment in patients with urticaria. Currently, the use of antihistamines has become popular due to its excellent safety profile and clinical efficacy, however to the investigators knowledge, there are no studies about the pharmacokinetic and pharmacodynamic effects of these drugs in patients of tropical Latin America. The investigators main interest is to evaluate if skin test inhibition correlates with the clinical effect of five anti-histamines.

DETAILED DESCRIPTION:
This was a randomized, double-blind, study that was conducted in six health care centers from Medellín and Bogotá (Colombia). This study was conducted in compliance with the ethical principles of the Declaration of Helsinki and with Good Clinical Practice guidelines. Written informed consent was obtained from all subjects or they parents in patients under 18 years. Ethical committee of University of Antioquia (Medellín, Colombia) approved the protocol. Considering the large number of articles that demonstrate the efficacy of antihistamines as first-line treatment in patients with urticaria, the ethics committee request that all participants would receive an antihistamine during the two months of the study because a placebo group would provide little information for the principal objective and the high risk of airway angioedema. Thirty heath subjects were used as a control group to evaluated the characteristics of the wheal in the prick test with histamine.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of persistent allergic urticaria.
* Age over 12 years and at least one year with the disease
* Informed consent filled.
* Be resident of the metropolitan area of Medellin.

Exclusion Criteria:

* • Use of immunosuppressive drugs

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with uticaria that improved Urticaria Activity Score and Life Quality Index (DLQI) with the use of antihistamine in mono-dose and quadruple dose. | Patients will be followed for two months
  Each patient will be assigned to receive the standard dose of one antihistamine for one month. The assignment of each patient group for each antihistamine will be using a double-blind system.
  In the second month, patients who do not achieve good control, will receive a quadrupled dose of the same antihistamine received in the first month.
  A medical evaluation, symptoms scales (UAS and DLQI) and prick test with histamine will be performed at enrollment and during the first and second months of follow up.

SECONDARY OUTCOMES:
Safety issue | 2 months
  Safety and tolerability were assessed by adverse events reported by subjects at each postrandomization clinic visit. We did electrocardiogram and laboratory examination before initiation of antihistamine therapy and each month after (complete blood count [CBC], aspartate aminotransferase [AST], alanine aminotransferase [ALT], creatinine, blood urea nitrogen). We did an specific questionnaire (in spanish) to assess sedation:
  "¿Sientes más sueño o somnolencia de lo acostumbrado?" (Do you feel more sleepy or drowsy than usual?), "¿Sientes que el sueño o la somnolencia interfiere con tus actividades diarias?" (Do you feel sleep or sleepiness interferes with your daily activities?), "¿Sientes que tú sueño no es reparador?" (Do you feel that you sleep is not restful?). Each question could be answered from 0 to 3 points (0 no 1. little, 2 moderate, 3 much). the sum of points defined them the severity of sedation in mild (0-3), moderate (4-5) and severe sedation (6-9).
Cholinergic and physical urticarias | 2 months
  We asked to each patients about physical triggers and with physical provocation test, we evaluated in all patients if wheals are evoked by a cholinergic or physical stimulus such as water, pressure, friction or cold contact.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Sánchez, M.D, Principal Investigator — IPS Universitaria, University of Antioquia
Locations (1):
- Medellin, Medellín, Antioquia, Colombia

REFERENCES:
- [Derived] Sanchez J, Zakzuk J, Cardona R. Evaluation of a Guidelines-Based Approach to the Treatment of Chronic Spontaneous Urticaria. J Allergy Clin Immunol Pract. 2018 Jan-Feb;6(1):177-182.e1. doi: 10.1016/j.jaip.2017.06.002. Epub 2017 Jul 12. PMID 28709817
- [Derived] Sanchez J, Zakzuk J, Cardona R. Prediction of the Efficacy of Antihistamines in Chronic Spontaneous Urticaria Based on Initial Suppression of the Histamine- Induced Wheal. J Investig Allergol Clin Immunol. 2016;26(3):177-84. doi: 10.18176/jiaci.0039. PMID 27326985